CLINICAL TRIAL: NCT06063551
Title: Cryopreservation of Prepubertal Testicular Tissue for Preservation
Brief Title: Cryopreservation of Prepubertal Testicular Tissue for Preservation of Fertility in Young Boys With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 140175
Record Dates: First submitted 2022-08-17; First posted 2023-10-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Fertility Disorders; Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The same protocol applies to all subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testicular Biopsy (Experimental): Patients meeting eligibility criteria are offered experimental procedure of testicular biopsy for clinical storage and use in laboratory research. The intervention does not involve a drug or device.
  Interventions: Procedure: Testicular Biopsy

INTERVENTIONS:
Procedure: Testicular Biopsy — Testicular biopsy for clinical storage and laboratory research.

SUMMARY:
Prepubertal boys treated for cancer are at risk of infertility as a result of their treatment. At present there are no options to preserve fertility in these boys. With informed consent, the investigators aim to cryopreserve (freeze) testis tissue biopsies taken from boys undergoing cancer therapy with a high risk of infertility. A portion of cryopreserved tissue will be securely stored, which in the future may be used to restore fertility in the patients. A second portion of the tissue will be used for laboratory work aimed at understanding the conditions required for development of the germ cells.

Patients will be recruited from the Oncology Department at the Royal Hospital for Children and Young People (RHCYP) in Edinburgh. Tissue will be obtained from prepubertal patients with cancer who are about to undergo treatment with a high risk (>80%) of infertility. Informed consent will be obtained from the patients legal guardian (and patient if applicable) for the procedure and subsequent use of tissue. A testis biopsy from one testis will be performed and if possible will coincide with a planned routine procedure requiring general anaesthetic in order to avoid the need for additional anaesthesia.

The procedure will take place at RHCYP during the initial assessment and prior to the commencement of cancer treatment and will not result in delay of treatment. Tissue will be assessed for the presence of sperm for storage using existing methods. In addition, tissue will be cryopreserved by Tissue and Cells Directorate, SNBTS in Edinburgh. The tissue will be stored for up to 55 years in accordance with current legislation (HFEA Act as amended 2005). Research will be carried out at the MRC Centre for Reproductive Health in accordance with Human Tissue (Scotland) Act 2006.

DETAILED DESCRIPTION:
Objectives

1. Primary Objective

   a) Cryopreservation of testicular tissue from pre- and peri-pubertal patients undergoing potentially sterilising therapy for future therapeutic use to preserve fertility.

   i. Development/refinement of inclusion and exclusion criteria ii. Exploration of patients and parents attitudes to this approach to fertility preservation iii. Development of the required multidisciplinary group to provide this
2. Secondary Objectives

   1. Follow-up patients after testis tissue cryopreservation
   2. Laboratory research - testicular germ cell development for fertility preservation i. Development of optimal freezing methods for testicular tissue ii. In-vitro culture methods for germ cell maturation iii. Development of xenografting approaches for maturation of germ cells

Design Prospective cohort study of pre- and peri-pubertal boys

Study Population Pre- and peri-pubertal boys due to undergo therapy with high risk of subsequent infertility

Main Study Endpoint Successful long-term cryostorage of testicular tissue for potential future use in fertility preservation, and follow-up of patients for effects of testicular biopsy on subsequent endocrine function

Establishment of laboratory techniques for the development of methods to support long term storage of tissue and methods for in vivo/in vitro spermatogenesis

Methods

Patient Recruitment Patients will be recruited from the Oncology Department at the RHCYP in Edinburgh. Testicular cryopreservation will be offered to eligible patients providing they meet the inclusion criteria. Age appropriate patient information sheets will be provided to the patients.

Patient Consent Consent will be for testis tissue cryopreservation and storage. Patients will also have the option of allowing tissue to be used for research purposes, however declining this aspect will not prevent them from consenting to cryopreservation of tissue. Due to the young age and immaturity of the study patients, written informed consent for a testicular biopsy under general anaesthetic will be obtained from the parents/guardian of the patient, unless the patients are considered able to give fully informed consent themselves. Patient assent will be sought from those boys not considered competent to provide written informed consent due to their young age.

Surgical Procedure The testicular biopsy will take place in operating theatres at the RHCYP before cancer gonadotoxic treatment begins. This will, whenever possible, coincide with a planned routine procedure requiring general anaesthetic in order to avoid the need for additional anaesthesia, hence this will not result in delay to commencing treatment. A blood sample will be taken for viral screening which is a requirement for tissue storage. The blood sample will be stored to allow further testing for infectious diseases as required over time by Tissues Services and the HTA.

Testicular volume will be assessed by visual inspection and manual palpation at surgery. The amount of tissue removed will typically be approximately 0.6-0.8mls from one testis, and never in excess of 50% of the total volume of a single testis. The procedure will involve a unilateral open testicular biopsy through a scrotal incision.

Since treatment with cytotoxic therapy will not have started prior to the biopsy, the risk of infection is minimal. In patients with solid tumours bleeding is unlikely to be a major problem since platelet numbers and function are generally normal in these patients. In patients with leukaemia thrombocytopenia is likely to be present at diagnosis, but haemostasis is routinely secured by platelet transfusion for operative procedures in these patients.

The biopsy will be taken for testis tissue cryopreservation, with a portion of the sample going for laboratory research (if consent has been obtained for this purpose). In pubertal patients, the tissue for cryopreservation will be immediately analysed by an experienced embryologist for the presence of sperm using standard methods. If sperm are present then a portion of the sample will be used for Testicular Sperm Extraction (TESE) and storage, whilst remaining tissue will be cryopreserved using methods described below.

Cryopreservation of testicular tissue Testis tissue will be stored under the licence terms of the HTA. Samples are collected into sterile Hank's balanced saline solution (HBSS; 14175-129; Life Technologies, Merelbeke, Belgium), and transported to Tissue Services for cryopreservation and storage.

1. Cryopreservation of Immature Testicular Tissue Cryopreservation of ITT is performed by placing two tissue pieces in each cryovial containing 0.7 M DMSO (D2650; Sigma-Aldrich, Bornem, Belgium), with 0.1 M sucrose (+S; 10274-5c; VWR, Leuven, Belgium) and 10 mg/ ml HSA as previously described (Keros, Hultenby et al. 2007) (Wyns, Curaba et al. 2007). Equilibration is performed at +4°C for 30 min. Using a programmable freezer, the vials are cooled at 1°C/min with holding at 0°C for 5 min, followed by cooling at 0.5°C/min until 20°C. At this temperature, the program is put on hold for 10 min to allow manual seeding. The program continues at a rate of 0.5°C/min until 240°C, held for 10 min, and continued to 270°C at 7°C/min, with subsequent plunging into liquid nitrogen.
2. Cryopreservation of Mature Testicular Tissue Each biopsy is minced carefully with two fine needles in a Petri dish with 2 mL HBSS or Human Tubule Fluid, supplemented with 2.5% HSA (adapted from Verheyen, De Croo et al. 1995). After centrifugation of the tissue/cell suspension at 500g for 10 min and removal of the supernatant, the pellet is resuspended in 200 µL HBSS or Human Tubule Fluid, supplemented with 2.5% HSA. SpermFreeze (Vitrolife) (is added slowly at a ratio of 1:1 (v/v) to the suspension. After 20 min of equilibration at 37°C, the sperm suspension is aspirated into a 500-µL cryostraw (IMV, l'Aigle Cedex, France). Cooling and freezing are carried out under computer control using a standard programme for ejaculated spermatozoa (Verheyen, Pletincx et al. 1993). The straws are placed into the chamber of a programmable biological freezer and cooled according to the following programme: (i) cooling rate of -1°C/min from room temperature to 4°C (ii) hold for 1 min (iii) freezing rate of -5°C/min from 4°C to -80°C (iv) plunge into liquid nitrogen (-196 °C).

Laboratory research The primary aim of this application is to store testis tissue from patients that may be used in the future for fertility preservation if required. However, consent will also be sought for use of an extra portion of tissue for laboratory research. In addition to obtaining tissue as described above, the investigators will also use tissues obtained from an alternative source of tissue obtained from a collaborating centre (John Radcliffe Hospital, Oxford, UK). This second source of human prepubertal testis material will be stored under a HTA licence (reference: 11106) in which consent has previously been obtained for the use of the tissue in approved research, including animal research.

This testis tissue will be used for three main aspects of laboratory research

1. Optimal freezing methods for pre-pubertal testis tissue and cells

   Freezing conditions need to be optimized and improved with xeno-free clinical grade components before clinical application can be considered. The investigators will assess the use of various cryoprotectants on survival and developmental potential of germ cells within the portion of pre-pubertal tissue taken for research. Post-thaw viability and functionality will be assessed by immunohistochemistry, flow cytometry and RT-PCR. To evaluate the functional properties of the tissue after freezing, the tissue will be xenografted or used for in-vitro culture.
2. In-vitro culture of pre-pubertal testis tissue

   Testis tissue organ culture using a soft agar system has resulted in full spermatogenesis using neonatal mouse testis (Sato, Katagiri et al. 2011). This method will be adapted for use with human pre-pubertal testis tissue by investigating the effects of different culture media, serum and the addition of gonadotrophins/other growth factors to stimulate germ cell differentiation. This will be evaluated by histological analysis and expression of markers for spermatogonia (e.g. MAGE-A4, Thy-1), spermatocytes (e.g. SCP-3, Prohibitin) and spermatids (e.g. Protamine-2, SP-10) which will be studied with different methodologies, including qPCR, flow cytometry and protein expression. Modifications of the culture conditions by adding the following substances will be considered: (1) Knock-out Serum Replacement (KO-SR) as it induced complete spermatogenesis in neonatal mouse testicular tissue culture (Sato, Katagiri et al. 2011); (2) Retinoic acid as it has a known role in meiosis and spermatogenic differentiation; (3) Testosterone as high concentrations of testosterone are essential for spermatogenesis in vivo.
3. Xenografting

Testis xenografting represents a model system to investigate the factors required to establish the spermatogonial stem cell (SSC) niche (Mitchell, Saunders et al. 2010). Testis tissue will be xenografted in mice, ectopically (dorsal skin, scrotal, kidney capsule) or directly into the testis in order to establish the SSC pool. The investigators will examine which factors are responsible for the maintenance of the SSC niche using established advanced immunohistochemical co-localisation studies. The investigators will determine protein expression in the SSCs and the surrounding niche, including somatic cells, basal lamina and vasculature. This will include proteins that have been shown to be important in SSC self-renewal/differentiation in rodents, such as c-kit/KITL and GDNF/Gfrα1. Grafts will also be maintained for longer periods in order to investigate subsequent differentiation of the germ cells beyond the spermatogonial stage by investigating morphology and expression of meiotic markers such as described for in-vitro work. The effects on the establishment of spermatogenesis by exposure of xenografts to exogenous gonadotrophins (LH/hCG +/- FSH) will also be determined. Moreover, the xenografting approach will be used to obtain SSCs which can then be propagated and/or transplanted into seminiferous tubules to achieve colonization.

Follow up of Patients Patients will be followed up in the Oncology clinic as normal until they are no longer required to have regular surveillance imaging when they will be transferred to the joint Oncology/Endocrinology 'Late Effects' clinic at the RHCYP in Edinburgh. Patients will be reviewed every 3 months through childhood and puberty to monitor growth and pubertal status. Subsequent follow up will be between 3 monthly and annually. Puberty will be assessed by clinical examination using Tanner Staging and also by measuring blood levels of gonadotrophins, testosterone and Inhibin B. Testicular volumes will be measured using a Prader orchidometer and an annual ultrasound of the testes will be performed to assess testicular growth and monitor for scarring or damage as a result of the biopsy. A key outcome is the prevalence of gonadal failure (divided into spermatogenic and endocrine) in boys who have had testicular biopsies in comparison with those with similar and other diagnoses who have not. This will ensure that in the unlikely event that there are adverse effects of the biopsy this will be detected and it will also allow modification of the selection criteria for biopsy and testis tissue cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and peripubertal boys
* Due to receive cancer treatment that is predicted to have a high risk (>80%) of infertility
* Consent to removal of testicular tissue for storage and research
* Unable to produce a semen sample by masturbation

Exclusion Criteria:

* Participation in study would delay treatment
* Too unwell to undergo the procedure
* Pre-existing testicular pathology/previous testicular surgery (eg orchidopexy)
* Able to produce a semen sample for cryopreservation

Ages: 1 Day to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Project is on male fertility and therefore by definition is only applicable to males. Similar programmes are already established for females.
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2061-04 (Estimated); Study Completion 2061-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of fertility | On reaching adulthood, typically 18 years.
  Semen analysis for sperm count
Reproductive hormones | On reaching adulthood, typically 18 years.
  Measurement of reproductive hormones in blood

SECONDARY OUTCOMES:
Germ Cell Development | 2 years
  Most advanced germ cell stage identified in tissue after culture or xenotransplant.

CONTACTS AND LOCATIONS:
Overall Officials: Rod T Mitchell, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No